CLINICAL TRIAL: NCT06232122
Title: Evaluation of 68Ga-FAPI-46 and 18F-FDG PET/CT Imaging for Detecting Recurrent Tumor Lesions in Patients of Ovarian Cancer With CA125 Elevation From Complete Response After Therapy
Brief Title: Evaluation of 68Ga-FAPI-46 and 18F-FDG PET/CT Imaging for Detecting Recurrent Tumor Lesions in Patients of Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Feng-Yuan Liu, MD, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202102208A0
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer
Keywords: 68Ga-FAPI-46; 18F-FDG; CA-125
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI ,PET/CT (Experimental): Inject 68Ga-FAPI and then perform PET/CT scan.
  Interventions: Diagnostic Test: 68Ga-FAPI-46; Diagnostic Test: 18F-FDG

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-46 — Intravenous injection of one dosage of 2 mCi 68Ga-FAPI-46
  Other Names: 68Ga-fibroblast activating protein inhibitors
Diagnostic Test: 18F-FDG — Intravenous injection of one dosage of 5-10mCi 18F-FDG
  Other Names: 18F-fluorodeoxyglucose

SUMMARY:
A prospective cohort imaging study in a single institution to evaluate 68Ga- FAPI-46 and 18F-FDG PET/CT imaging for detecting recurrent tumor lesions in patients of ovarian cancer with CA125 elevation from complete response after therapy

DETAILED DESCRIPTION:
Ovarian cancer is the eighth most common cancer worldwide in females and usually diagnosed at an advanced stage. Serum cancer antigen 125 (CA125) is widely used in ovarian cancer. An elevation in CA125 levels can precede a clinically apparent recurrence by 3 to 6 months and 18F-FDG PET/CT can modify management in approximately half of these patients. However. 18F-FDG PET/CT may yield false negative results. 68Ga-FAPI-46 PET/CT shows potential here. This study is to assess the diagnostic performances of 68Ga-FAPI-46 and 18F-FDG PET/CT for ovarian cancer recurrence in patients with CA125 elevation from complete response after therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven ovarian cancer with complete response after therapy
* Age between 30 and 80
* Elevation of serum CA125 value above the normal range (>35 U/mL) or doubling of serum CA125 value within the normal range
* ECOG performance status grade 0 or 1 and willing to receive further therapy if disease recurrence is confirmed
* Willing to enter this prospective study with signed informed consent form

Exclusion Criteria:

* Patients with history of other malignancy
* Patients who are pregnant or lactating
* Patients with fasting fingerstick glucose level higher than 200 mg/dl
* Known allergic reactions to components of the radiopharmaceutical solutions for intravenous injection for 68Ga-FAPI-46 or 18F-FDG imaging studies
* Patients who are incapable of lying still for 30 minutes to receive the PET/CT scan as assessed by investigators

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performances of 68Ga-FAPI and 18F-FDG PET/CT for ovarian cancer recurrence after one year from PET/CT imaging in Per-Protocol Analysis Dataset | 2 months for individual participants to complete all visits
  Diagnostic performance is defined as the AUC value of ROC curve (sensitivity against 1-specificity at different PET/CT imaging scores ranged from 1 to 4).
  Cancer recurrence is defined by pathological or imaging evidence up to one year after 68Ga-FAPI-46 PET/CT study.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 5 years
  Progression-free survival (PFS) is defined as the duration (months) from the initiation of further therapy to disease progression assessed by Gynecological Cancer Intergroup (GCIG) guideline which incorporates both RECIST 1.1 and CA125 or to death.
Overall Survival (OS) | 5 years
  Overall survival (OS) is defined as the duration (months) from the 68Ga-FAPI-46 PET/CT study to death.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang-Gung Memorial Hospital, Linkou Branch, Taoyuan, Taiwan